CLINICAL TRIAL: NCT02702921
Title: A Prospective, Randomized, Controlled, Multi-Center Evaluation of a Powered Vascular Stapler in VAT Lobectomies
Brief Title: Powered Vascular Stapler in Video-Assisted Thoracoscopic (VAT) Lobectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESC-15-001
Record Dates: First submitted 2016-03-02; First posted 2016-03-09 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgeon's 'standard of care' stapler (Active Comparator): Surgeon's current standard of care stapler
  Interventions: Device: Surgeon's 'standard of care' stapler
- Ethicon Powered Vascular Stapler (Experimental): Ethicon Powered Vascular Stapler
  Interventions: Device: Ethicon Powered Vascular Stapler

INTERVENTIONS:
Device: Surgeon's 'standard of care' stapler
  Arms: Surgeon's 'standard of care' stapler
Device: Ethicon Powered Vascular Stapler
  Arms: Ethicon Powered Vascular Stapler

SUMMARY:
This prospective, randomized, controlled, multi-center study will collect and compare data from the surgeon's current Standard Of Care stapler (for Pulmonary Artery/Pulmonary Vein transection) and powered vascular stapler.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed or suspected diagnosis of stage IA to stage IIIA non-small cell lung cancer scheduled for a lobectomy (Lung Cancer Staging per American Joint Committee on Cancer,7th Edition)5;
* Subjects scheduled for VATS lobectomy in accordance with their institution's Standard Of Care;
* Performance status 0-1 (Eastern Cooperative Oncology Group classification);
* American Society of Anesthesiologists (ASA) score </= 3;
* No prior history of VAT or open lung surgery (on the lung in which the procedure will be performed);
* Willing to give consent and comply with study-related evaluation and treatment schedule; and
* At least 18 years of age.

Exclusion Criteria

* Prior chemotherapy or radiation (within 30 days prior to the procedure or the duration of the subject's enrollment);
* Pregnancy;
* Physical or psychological condition which would impair study participation; or
* The subject is judged unsuitable for study participation by the Investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=11732&filename=ESC-15-001%20Protocol%20FINAL%20with%20NCT%20ID.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=11732&filename=ESC-15-001%20Final%20Protocol%20VATS%2011NOV2015_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from Feb 2016 to Feb 2017 across 7 hospitals.
Pre-assignment Details: 229 subjects signed an informed consent, 201 were randomized into one of the two groups. The 28 not randomized did not meet the inclusion criteria.
Groups:
- Standard of Care: Facility's Current Instrumentation
- Powered Vascular Stapler: Use of the ECHELON FLEX™ Powered Vascular Stapler
Period: Overall Study
Arm/Group | Standard of Care | Powered Vascular Stapler
Started (February 2017) | 98 | 103
Completed (March 2017) | 84 | 95
Not Completed | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Powered Vascular Stapler | Total
Number analyzed (Participants) | 98 | 103 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participant Age in Years
  Years | 68.2 (9.1) | 68.0 (9.0) | 68.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 60 | 105
  Male | 53 | 43 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 25
  Not Hispanic or Latino | 66 | 70 | 136
  Unknown or Not Reported | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 94 | 98 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Intra-Operative Hemostatic Intervention
Description: Incidence of hemostatic interventions/procedures completed for intra-operative bleeding related to the transection of the Pulmonary Artery and Pulmonary Vein during Video Assisted Thoracoscopic lobectomy with the use of standard of care stapler (SOC) or powered vascular stapler (PVS) defined as bleeding detected and controlled intraoperatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurs intra-operatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open).
Time Frame: Intra-Operative, an average of 2.3 hours, ranging from 30 mintues to 6.4 hours
Population: A total of 229 subjects were screened and 201 subjects were randomized into the study - 98 randomized to SOC and 103 randomized to PVS. Two subjects randomized to SOC stapler received the PVS group. These subjects are included in the stapler group for the primary endpoint analysis, consistent with the intention-to-treat principle.
Measure: Number (95% Confidence Interval); unit: Proportion transections w/ intervention
Units Other Than Participants: Vessels Transection
Arm/Group | Standard of Care | Powered Vascular Stapler
Number analyzed (Participants) | 98 | 103
Number analyzed (Vessels Transection) | 300 | 336
Proportion transections w/ intervention | 0.0533 [0.0279 to 0.0788] | 0.0833 [0.0538 to 0.1129]

2. Secondary Outcome: Post-operative Interventions or Procedures Related to Pulmonary Artery or Pulmonary Vein Bleeding
Description: Incidence of hemostatic interventions /procedures completed for post-operative bleeding related to the transection of the PA and PV during VATS lobectomy with the use of SOC or PVS:
  * Hemostasis intervention: bleeding that occurs post-operatively requiring blood or blood product transfusion or an additional surgical procedure (related to PA and PV transection).
  No hemostasis intervention is defined as no interventions needed for post-operative bleeding (related to PA and PV transection).
Time Frame: Post-Op through 4 Week Followup
Population: A total of 229 subjects were screened and 201 subjects were randomized into the study - 98 randomized to SOC and 103 randomized to PVS. Two subjects randomized to SOC stapler received the PVS stapler. These subjects are included in the PVS group for safety analysis.
Measure: Number (95% Confidence Interval); unit: Proportion participants w/ intervention
Units Other Than Participants: Participant
Arm/Group | Standard of Care | Powered Vascular Stapler
Number analyzed (Participants) | 96 | 105
Number analyzed (Participant) | 96 | 105
Proportion participants w/ intervention | 0.0104 [0.0000 to 0.0307] | 0.0095 [0.0000 to 0.0281]

ADVERSE EVENTS:
Time Frame: 4 Weeks Post Procedure
Description: For safety reporting, subjects are counted under the device that was actually used. For Participant Flow, Baseline and Outcome Measures, subjects are counted in their randomized group consistent with the intention-to-treat principle. Two subjects who were randomized to Standard of Care were operated on with the Powered Vascular Stapler (PVS), thus these 2 are counted in the PVS group for Adverse Event summaries, thus the difference in total number at risk when comparing to the Participant Flow.
Arm/Group | Standard of Care | Powered Vascular Stapler
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/105
Serious Adverse Events (participants affected / at risk) | 22/96 | 18/105
Other Adverse Events (participants affected / at risk) | 35/96 | 33/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=96) | Powered Vascular Stapler (N=105)
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Infarction (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=96) | Powered Vascular Stapler (N=105)
Atrial fibrillation (Cardiac disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 3 | 1
Pain (General disorders) | 1 | 4
Pneumonia (Infections and infestations) | 5 | 3
Wound infection (Infections and infestations) | 4 | 0
Arterial injury (Injury, poisoning and procedural complications) | 3 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 6
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT02702921/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02702921/SAP_001.pdf